CLINICAL TRIAL: NCT06457776
Title: Medication Related Osteonecrosis of the Jaws (MRONJ) in a Cohort of Patients Treated by Antiresorptive Drugs: a Cohort Prospective Study
Brief Title: Medication Related Osteonecrosis of the Jaws (MRONJ) in a Cohort of Patients Treated by Antiresorptive Drugs
Status: Recruiting | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Lajolo, Associate Professor, Catholic University of the Sacred Heart
Other Study IDs: MRONJ-1
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Osteonecrosis of the Jaw; Osteonecrosis Due to Drugs, Jaw; Osteonecrosis Due to Drug; Bisphosphonate-Associated Osteonecrosis; Bisphosphonate-Associated Osteonecrosis of the Jaw
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw | interventions — Practice Management, Dental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antiresorptive Drugs: Patients treated by means of Antiresorptive drugs due to either bone metastasis or metabolic diseases
  Interventions: Procedure: Dental management

INTERVENTIONS:
Procedure: Dental management — The oral conditions of the included patients will be evaluated at baseline. When indicated, dental extractions will be performed before the beginning of Antiresorptive Therapy. Patients will then receive a six-months intervals follow-up, during which primary and secondary prevention of dental diseases will be performed.

SUMMARY:
The objective of this prospective observational study is to investigate the incidence of Medication Related Osteonecrosis of the Jaws (MRONJ) in patients receiving antiresorptive drugs for oncohematologic reasons during a 5-year follow-up. Secondary objectives are to compare the different antiresorptive drugs in relation to the incidence of MRONJ and to identify any systemic as well as local risk factors.

DETAILED DESCRIPTION:
Antiresorptive drugs are widely used for the prevention and treatment of numerous diseases involving the skeletal system. In particular, they have been shown to be effective in reducing the incidence of skeletal events in oncohematologic patients.

Specifically, bone represents a highly affected site of metastatic cancer (i.e., bone metastases from solid tumors of various origins--breast, prostate, renal; multiple myeloma). In the United States, approximately 400,000 individuals suffer from bone metastasis. The most frequent skeletal complications in patients with bone metastases (referred to as SRE - skeletal-related events - in the international literature) include pathologic fractures, spinal cord compression, malignant hypercalcemia, and the need to undergo radiation therapy or surgery on the bone lesion.The introduction of anti-bone resorption drugs (bisphosphonates and denosumab) has reduced the rate of skeletal complications by 30-50% so they are indicated in the management of the oncohematology patient.

The objective of this prospective observational study is to investigate the incidence of Medication Related Osteonecrosis of the Jaws (MRONJ) in patients receiving antiresorptive drugs for oncohematologic reasons during a 5-year follow-up. Secondary objectives are to compare the different antiresorptive drugs in relation to the incidence of MRONJ and to identify any systemic as well as local risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with specific prescription to initiate therapy with antiresorptive drugs

Exclusion Criteria:

* Previous Head and Neck Radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients starting an antiresorptive drug
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Medication Related OsteoNecrosis of the Jaws | Five years after the beginning of AR therapy
  Incidence of Medication Related OsteoNecrosis of the Jaws

CONTACTS AND LOCATIONS:
Locations (1):
- Cosimo Rupe, Roma, Italy